CLINICAL TRIAL: NCT01107756
Title: A Phase IV Clinical Trial of Patients With Solid Tumours Receiving Granocyte 34 (Granulocyte Colony Stimulating Factor (G-CSF)) as Primary Prophylaxis for Chemotherapy-induced Neutropenia, in a Taxotere (Docetaxel) Based Regimen
Brief Title: A Clinical Trial of Patients With Solid Tumours Receiving Granulocyte Colony Stimulating Factor as Primary Prophylaxis for Chemotherapy-induced Neutropenia, in a Docetaxel Based Regimen
Acronym: Grano-Tax
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_04775; U1111-1116-9574 (Other: UTN)
Record Dates: First submitted 2010-04-13; First posted 2010-04-21 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Neoplasms (no Otherwise Specified)
MeSH Terms: conditions — Neoplasms | interventions — Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAXOTERE (Docetaxel) + GRANOGYTE 34 (Lenograstim) (Experimental): Taxotere (Docetaxel) is given as background treatment and should be administered by the treating physician in accordance with the prescribing information outlined in the package insert + Granocyte 34 (lenograstim)
  Interventions: Drug: LENOGRASTIM (GRANOGYTE 34)

INTERVENTIONS:
Drug: LENOGRASTIM (GRANOGYTE 34) — Pharmaceutical form: solution Route of administration: intravenous Dose regimen:recommended dosing as per Granocyte 34 package insert

SUMMARY:
Primary Objective:

To evaluate the incidence and severity of neutropenia in patients being treated for solid tumours with a Taxotere® based regimen when Granocyte® 34 is being used as a primary prophylaxis for chemotherapy-induced neutropenia.

Secondary Objectives:

Haematological : To evaluate the incidence and severity of febrile neutropenia (with or without antibiotics) and anaemia in patients being treated for solid tumors treated with a Taxotere based regimen when Granocyte is being used as a primary prophylaxis.

Non-Haematological : To evaluate the incidence and severity of the following adverse events: asthenia, anorexia, myalgia, nail changes and oral mucositis in patients with solid tumours treated with a Taxotere based regimen; when Granocyte is being used as a primary prophylaxis.

ELIGIBILITY:
Inclusion criteria:

* Patients willing to sign informed consent prior to entry into the study,
* Patients who have been prescribed a Taxotere based regimen,
* Patients who have not yet started with the first Taxotere treatment,
* Patients with a histological diagnosis of one of the following solid tumours: breast cancer, non-small cell lung cancer (NSCLC), ovarian cancer, prostate cancer, gastric cancer or head and neck cancer.

Exclusion criteria:

* Patients who are enrolled in another clinical study,
* Pregnant and/or breastfeeding patients, including women of childbearing potential not willing to use medically acceptable methods of contraception,
* Patients with severe liver impairment,
* Patients with severe renal function impairment,
* Patients with a known hypersensitivity to Granocyte 34 or its constituents,
* Patients with a history of severe hypersensitivity reactions to Taxotere or Polysorbate 80,
* Patients with a baseline neutrophil count of < 1500cells/mm3,
* Patients on other drugs that are contra-indications for the use with Taxotere,
* Patients on con-current radiotherapy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of neutropenia assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4. | For each granocyte 34 treatment, from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal

SECONDARY OUTCOMES:
Incidence and severity of febrile neutropenia assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence and severity of anaemia assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence and severity of asthenia assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence and severity of anorexia assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence and severity of myalgia assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence and severity of nails changes, including nail disorders assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence and severity of oral mucositis assessed by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Neutropenia/febrile neutropenia associated days in hospital | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Neutropenia/febrile neutropenia associated use of anti-infectives | for each granocyte 34 treatment from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Incidence of chemotherapy dose reduction, withdrawals or treatment delays due to neutropenia or febrile neutropenia | from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Infection with (or without) neutropenia | from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal
Relationship between the incidence and severity of neutropenia and the different chemotherapy regimens | from the the study start (visit 1) to the study end (Follow-up visit at 30 (±9) days post Taxotere treatment or with premature withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- South Africa (25):
  - Investigational Site Number 53, Alberton
  - Investigational Site Number 55, Benoni
  - Investigational Site Number 11, Bloemfontein
  - Investigational Site Number 21, Cape Town
  - Investigational Site Number 27, Cape Town
  - Investigational Site Number 26, Cape Town
  - Investigational Site Number 22, Cape Town
  - Investigational Site Number 13, Durban
  - Investigational Site Number 14, Durban
  - Investigational Site Number 32, East London
  - Investigational Site Number 012, eManzimtoti
  - Investigational Site Number 24, George
  - Investigational Site Number 51, Johannesburg
  - Investigational Site Number 12387, Johannesburg
  - Investigational Site Number 47, Klerksdorp
  - Investigational Site Number 43, Mbombela
  - Investigational Site Number 44, Polokwane
  - Investigational Site Number 31, Port Elizabeth
  - Investigational Site Number 42, Pretoria
  - Investigational Site Number 41, Pretoria
  - Investigational Site Number 451, Pretoria
  - Investigational Site Number 48, Rustenburg
  - Investigational Site Number 54, Sandton
  - Investigational Site Number 25, Somerset West
  - Investigational Site Number 56, Vereeniging